CLINICAL TRIAL: NCT02197143
Title: A Comparison of Efficacy of Intravenous Esomeprazole and Ranitidine Treatment of Dyspeptic Pain: A Double-Blind, Randomized, Controlled Trial
Brief Title: A Comparison of Efficacy of Intravenous Esomeprazole and Ranitidine Treatment of Dyspeptic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, hayri elicabuk, md, Pamukkale University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MDhayri84; 120841 (Other: Drug and Medical Device Institution)
Record Dates: First submitted 2014-07-09; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Dyspepsia
Keywords: esomeprazole; ranitidine; hydrotalcid; treatment of dyspepsia; emergancy medicine
MeSH Terms: conditions — Dyspepsia | interventions — Esomeprazole; Ranitidine; hydrotalcite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Esomeprazole (Experimental): 40 mg Esomeprazole in 150 ml normal saline given as a slow intravenous infusion over 15 minutes and p.o. 10ml Hydrotalcid
  Interventions: Drug: esomeprazole; Drug: hydrotalcid
- Ranitidine (Experimental): 50mg Ranitidine in 150 ml normal saline given as a slow intravenous infusion over 15 minutes and p.o. 10ml Hydrotalcid
  Interventions: Drug: esomeprazole; Drug: Ranitidine
- placebo (Experimental): 150 ml only normal saline given as a slow intravenous infusion over 15 minutes and p.o. 10ml Hydrotalcid
  Interventions: Drug: Ranitidine; Drug: hydrotalcid

INTERVENTIONS:
Drug: esomeprazole — 40 mg esomeprazole in 150 ml normal saline given as a slow intravenous infusion over 15 minutes and p.o. 10ml Hydrotalcid
  Other Names: Nexium, Astra Zeneca drugs, Södertalje; Esmara; Esom
  Arms: Esomeprazole; Ranitidine
Drug: Ranitidine — 50mg Ranitidine in 150 ml normal saline given as a slow intravenous infusion over 15 minutes and p.o. 10ml Hydrotalcid
  Other Names: Ulcuran, Abfar drugs, Istanbul; Ranitab; Ultidin
  Arms: Ranitidine; placebo
Drug: hydrotalcid — 150 ml only normal saline given as a slow intravenous infusion over 15 minutes and p.o. 10ml Hydrotalcid
  Other Names: Talcid, Bayer, Istanbul
  Arms: Esomeprazole; placebo

SUMMARY:
* Currently, Proton Pump Inhibitors and H2Receptor Blockers are widely used by emergency physicians in Turkey for the treatment of patients with dyspepsia.
* The objective of the study was to assess whether intravenous esomeprazol has superior dyspeptic pain reduction compared with ranitidine or hydrotalcid in emergency department (ED) adults
* The investigators second aim was to compare recurrent dyspeptic pain within 24 hours after discharge and cost of treatments in the treatment of dyspepsia.

DETAILED DESCRIPTION:
* this is the placebo randomized double blinded clinical trial to compare the efficacy of these three drugs in this clinical setting.
* A randomized clinical trial was conducted in the ED of Pamukkale University Medical Faculty Hospital
* Study personnel (emergency physicians and nurses) were trained before the study.
* When intravenous drugs (esomeprazol, ranitidine or plasebo) was being recommended, an eligibility checklist was completed by the attending physician.
* If there were no exclusion criteria, written informed consent was obtained and baseline information, including initial dispeptic pain severity ratings with VAS were recorded.
* The need for identification and enrollment of participants by staff with conflicting work pressures resulted in recruitment of a convenience sample of patients.
* All patients eligible for the study were randomized to one of three groups:
* First Group: 40 mg Esomeprozol with 5 cc syringe in 150 ml normal saline given as a slow intravenous infusion over 15 minutes and p.o. 10ml Hidrotalcid
* Second Group: 50mg Ranitidin with 5 cc syringe in 150 ml normal saline given as a slow intravenous infusion over 15 minutes and p.o. 10ml Hidrotalcid
* Third Group: 150 ml only normal saline given as a slow intravenous infusion over 15 minutes and p.o. 10ml Hidrotalcid
* Drug packs prepared in 5 ml syringes were numbered by an independent nurse, who not involved in the study.
* Drug packs were prepared according to the computer-generated random number sequence to assign treatment allocations
* The allocation list was kept by the emergency nurse. Patients received the esomeprazol, the ranitidin or the placebo medication schemes according to their random allocations.
* After enrollment and recording of baseline information, the next numbered study drug pack was obtained, and administered as a infusion over 15 minutes.
* Randomization was achieved by using computer software to generate random numbers. During the intervention, participants were monitored by an oxygen saturation (SpO2) monitor, an automatic sphygmomanometer (blood pressure), and a rhythm monitor (heart rate and rhythms)
* One researcher blinded to patient allocation observed the whole procedure and recorded the dyspeptic pain scores.
* Patients in both groups received three types of medication in a similar manner (for example, 150 ml normal saline given as a slow intravenous infusion over 15 minutes), thus ensuring double blinding.
* Dyspeptic pain scores were recorded at 0, 15, 30, 45 and 60 min on a VAS of 1 to 10
* Rescue medication [hidrotalcid 10ml (Talcid, Bayer, Istanbul, Turkey)] was given intravenously to patients if dyspeptic pain VAS scores ≥ 5 in thirty minutes after study drug administration.
* All other medications required during the study also were recorded.
* During the study, pulse rate, systolic blood pressure, diastolic blood pressure, respiration rate and oxygen saturation (SpO2) were recorded at baseline (0 min), 15, 30, and 60 min.

ELIGIBILITY:
Inclusion Criteria:

* patients were eligible for inclusion if they were aged 18 years or older, 60 years or older,
* had dyspspsia [VAS (visual analog scale) score >5] during their ED episode of care for which the attending physician recommended medication.

Exclusion Criteria:

* pretreatment 100-mm linear visual analog scale (VAS) pain score less than 50 mm;
* known cases of malignancy or terminal illness;
* known cases of major medical problems (eg, any evidence of active structural or functional abnormality of the hearts, chronic renal failure)
* allergy or previous adverse reaction to study drugs studied
* received agents to inhibit the secretion of acid (PPIs or histamine-2 receptor antagonists), nonsteroidal anti-inflammatory drugs,
* who consumed alcohol within 4 hours before the ED visit
* diarrhea more than 2 times within the past 24 hours;
* being suspected to have other ED diagnoses (eg, gut obstruction, biliary colic, pancreatitis, hepatitis, or localized hepatobiliary infections);
* being pregnant or breast-feeding; and
* inability to comprehend the VAS evaluation.
* and patients who refused to participate study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 286 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
compare the effects of intravenous esomeprazol and ranitidin for the treatment of dyspepsia in the emergency setting. | Patients in both groups received three types of medication than dyspeptic pain scores were recorded at 0, 15, 30, 45 and 60 min on a VAS of 1 to 10.
  This work took 17 months

CONTACTS AND LOCATIONS:
Overall Officials: hayri elicabuk, md, Principal Investigator — pamukkale universty
Locations (1):
- Pamukkale Universty, Denizli, Denizli, Turkey (Türkiye)